CLINICAL TRIAL: NCT06594367
Title: A Possible Founding PKD2 Mutation Associated With Variable Phenotypes of ADPKD in Bergamo Province
Acronym: POPULAR
Status: Active, not recruiting | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: POPULAR
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Keywords: PKD2 mutation; founder effect; Bergamo province; variable phenotype
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: 10 patients from di 7 families living in 3 villages of the Bergamo province i.e., Torre de Roveri, Albano S. Alessandro and Scanzorosciate who during genetic tests for ADPKD have revealed the presence of a new heterozygous deletion in the PKD2 gene will be included in this study.

SUMMARY:
This is an observational study aimed at assessing if a new and specific heterozygous deletion detected at PKD2 gene is associated to a "founder effect" in 10 Autosomal dominant polycystic kidney disease (ADPKD) patients, and at investigating the genotype-phenotype correlation in the families sharing the same PKD2 breakpoint site.

DETAILED DESCRIPTION:
Autosomal dominant polycystic kidney disease (ADPKD) is the most common inherited disease of the kidney. It occurs in adulthood but is also rarely diagnosed in early childhood. The majority of the disease-causing variants observed in ADPKD patients are located in two genes: PKD1 and PKD2. They account for 78% and 13% of ADPKD cases, respectively, while in approximately 6-9% of clinically diagnosed patients other genes have been shown to contribute to the disease.

Most ADPKD mutations are private and so far no hot-spot mutations have been reported in PKD1 and PKD2. On average, renal survival of patients with PKD2 mutations is 20 years longer than in patients with PKD1 mutations. However, there is a high degree of clinical variability among patients as well as within families, with different rates of progression towards end-stage renal disease (ESRD), partially driven by genetic factors.

Few reports are available about possible founding mutations in ADPKD. We have recently reported the results of genetic analysis for PKD1 and PKD2 by Sanger sequencing and Multiplex Ligation-dependent Probe Amplification (MLPA) in a large Italian cohort of ADPKD patients who were referred to our center for genetic analysis through the Italian National Health Service.

MLPA is a method for detecting copy number variation (CNV) of a specific DNA segment within the genome, suggestive of duplications, deletions or other structural variants that may affect long DNA stretches. The exact characterization of the extent of the structural variant identified by MLPA, however, requires subsequent analyses.

In 4 families (6 patients) who were negative at Sanger sequencing, MLPA analysis of PKD2 revealed a novel heterozygous copy number variation (CNV) indicative of a deletion of at least 11,000 base pairs (bp) and spanning exons 1-2. These families are formally not related, but they live in the same geographical area including three small villages in Bergamo province (Torre de Roveri, Albano S. Alessandro, Scanzorosciate), suggesting a potential founder effect. More recently, we detected the same PKD2 CNV in 3 additional families (4 patients) from the same geographical area, further strengthening this hypothesis. Most affected subjects in these families have mild disease, as expected for PKD2 mutations, but one patient experienced early ESRD and another one presents congenital anomalies of the kidney and the urinary tract (CAKUT) in addition to the typical ADPKD phenotype, indicating a different expressivity of the disease or the possible presence of other genetic factors affecting the clinical phenotype.

Further in depth analyses were needed to investigate the deletion of at least 11,000 base pairs (bp) and spanning exons 1-2 to find the breakpoint site in the 10 patients for diagnostic purpose. We found the same breakpoint sites across all the patients pointing to a common origin, and similar disease expressivity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ADPKD

Exclusion Criteria:

* Healthy patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Italian cohort of ADPKD patients who were referred to the Clinical Research Centre for Rare Diseases Aldo e Cele Daccò for genetic analysis through the Italian National Health Service.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-10-12 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Evidence of a deletion | At day 1
  Evidence of an heterozygous copy number variation (CNV) indicative of a deletion of at least 11,000 base pairs (bp) and spanning exons 1-2 (DNA amplification by long-range PCR).
Genetic counseling | At day 1
  All the patients sharing the same PKD2 deletion will be interviewed about their personal and familial anamnesis. Starting from the pedigree and the detailed family medical history, the genotype-phenotype correlation will be defined and other potentially affected family members, if any, will be identified.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Centre for Rare Diseases Aldo e Cele Daccò, Ranica, BG, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Orisio S, Noris M, Rigoldi M, Bresin E, Perico N, Trillini M, Donadelli R, Perna A, Benigni A, Remuzzi G. Mutation Analysis of PKD1 and PKD2 Genes in a Large Italian Cohort Reveals Novel Pathogenic Variants Including a Novel Complex Rearrangement. Nephron. 2024;148(5):273-291. doi: 10.1159/000530657. Epub 2023 May 25. PMID 37231942
- [Background] Willey CJ, Blais JD, Hall AK, Krasa HB, Makin AJ, Czerwiec FS. Prevalence of autosomal dominant polycystic kidney disease in the European Union. Nephrol Dial Transplant. 2017 Aug 1;32(8):1356-1363. doi: 10.1093/ndt/gfw240. PMID 27325254
- [Background] Cornec-Le Gall E, Audrezet MP, Chen JM, Hourmant M, Morin MP, Perrichot R, Charasse C, Whebe B, Renaudineau E, Jousset P, Guillodo MP, Grall-Jezequel A, Saliou P, Ferec C, Le Meur Y. Type of PKD1 mutation influences renal outcome in ADPKD. J Am Soc Nephrol. 2013 May;24(6):1006-13. doi: 10.1681/ASN.2012070650. Epub 2013 Feb 21. PMID 23431072